CLINICAL TRIAL: NCT07324109
Title: Clinical Application Observation: Evaluation of Phantom Limb Pain After 3 Weeks of Use of a Feedback System Using Vibration (Suralis, Manufacturer: Saphenus)
Brief Title: Clinical Application Observation on the Evaluation of Phantom Limb Pain With the Suralis System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Median (Other)
Responsible Party: Principal Investigator, Johannes Schroeter, Dr. med. Johannes Schroeter, Median
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PhantomLimbPain
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Phantom Limb Pain After Amputation; Lower Limb Amputation Above Knee; Lower Limb Amputation Below Knee; Lower Limb Amputation Knee
Keywords: Phantom limb pain; Vibrotactile feedback; Lower limb amputation; Suralis system; Pain management
MeSH Terms: conditions — Phantom Limb; Agnosia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention with Suralis System (Experimental): All participants receive a 3-week intervention with the Suralis vibrotactile feedback system, which provides real-time pressure-based sensory feedback via a sensorized insole and thigh-mounted vibrating cuff, calibrated individually via smartphone app to support pain reduction and gait stability.
  Interventions: Device: Vibrotactile sensory feedback

INTERVENTIONS:
Device: Vibrotactile sensory feedback — The Suralis system delivers real-time vibrotactile feedback via four pressure sensors embedded in a prosthetic insole, each mapped to a corresponding vibration motor on a thigh cuff. Participants wear the device during daily ambulation for 3 weeks. Vibration parameters (threshold, intensity, duration, spatial mapping) are individually calibrated via a smartphone app to match each user's sensory perception and gait pattern. The system operates autonomously, requires daily charging, and logs usage data via Bluetooth. No additional therapy or medication is administered alongside the device. The intervention aims to modulate cortical reorganization and reduce phantom limb pain while improving gait confidence and safety, particularly under non-visual conditions (e.g., stepping backward or sideways). The device is CE-marked (UDI: FBS 1 912012142) and classified as a Class IIa medical device under EU MDR 2017/746.

SUMMARY:
This study tests whether a vibration-based feedback device (Suralis) can reduce phantom limb pain in people with lower-leg amputations over 3 weeks. Participants wear the device daily and report pain levels, walking ability, and quality of life - with no known risks, as it's a CE-certified medical device. If pain improves, the study team will help participants apply for insurance coverage to keep using the system long-term. The goal is to offer a simple, non-drug option that may help ease chronic pain and improve daily function for amputees. Participation is voluntary and can be stopped anytime without affecting medical care.

DETAILED DESCRIPTION:
This observational, prospective, single-arm pilot study evaluates the short-term effects of the Suralis vibrotactile feedback system (Saphenus Medical Technology GmbH) on phantom limb pain intensity, gait stability, and perceived quality of life in individuals with unilateral lower-limb amputation. The Suralis system consists of a sensorized insole with four pressure-sensitive zones (toe, forefoot, midfoot, heel), each mapped to a corresponding vibrotactile actuator embedded in a thigh-mounted cuff. Vibration parameters - including onset threshold, intensity (0-100 % amplitude), duration (50-500 ms), and spatial mapping - are individually calibrated via a proprietary iOS/Android app, allowing for personalized somatosensory substitution. The system operates autonomously during ambulation.

The study protocol includes a 3-week baseline phase to confirm persistent phantom pain (VAS ≥ 3/10 daily), followed by 3 weeks of active intervention, and a 3-week washout/follow-up phase to assess sustainability of effects. All assessments are conducted at the study center and include standardized functional tests (TUG, 6MWT), validated German-language questionnaires (DSF, VR-12, DASS, FW7, GCPS), and daily VAS entries captured via paper-based diaries. The system's CE-marked status (UDI: FBS 1 912012142) confirms conformity with EU MDR 2017/746 for Class IIa medical devices; no adverse events related to device use have been reported in prior clinical use. The study design incorporates no control group or randomization, reflecting its exploratory, real-world application focus. Statistical analysis will be descriptive and exploratory, with non-parametric methods applied to ordinal outcomes (Friedman test) and parametric or non-parametric repeated-measures analyses for continuous variables, depending on distribution. No blinding is feasible due to the nature of the intervention. All procedures comply with the Declaration of Helsinki and have been reviewed by the Ethics Committee of the Hessian Medical Association (approval pending).

ELIGIBILITY:
Inclusion Criteria:

* Unilateral major lower-limb amputation (transtibial or transfemoral)
* Presence of persistent phantom limb pain, defined as daily pain intensity ≥ 3/10 on the Visual Analog Scale (VAS) during the baseline period
* Regular daily use of a prosthetic limb (minimum 4 hours/day)
* Adequate German language proficiency to understand and complete study questionnaires and follow study procedures
* Ability to provide informed consent

Exclusion Criteria:

* Unstable wound or skin condition at the residual limb
* Inconsistent prosthetic use (less than daily or < 4 hours/day)
* Poorly fitting or non-functional prosthesis (as determined by study team)
* Incapacity to provide informed consent (e.g., due to cognitive impairment or severe psychiatric illness)
* Insufficient German language skills to comprehend study materials or complete assessments reliably

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Baseline (t1), end of 3-week intervention (t3), and 3-week follow-up (t4) - assessed via daily VAS entries averaged per time point.
  Scores range from 0 to 100 mm, where 0 mm = "no phantom pain" and 100 mm = "worst imaginable phantom pain"; higher scores indicate greater pain intensity.

SECONDARY OUTCOMES:
German Pain Questionnaire DSF - subscales | Baseline (t1), end of 3-week intervention (t3), and 3-week follow-up (t4) - completed in person at study center.
  A validated, German-language questionnaire that captures pain intensity, quality, chronicity (GCPS), well-being (FW7), psychological status (DASS) and health-related quality of life (VR-12).
Timed Up-and-Go (TUG) test | Baseline (t1), end of 3-week intervention (t3), and 3-week follow-up (t4) - performed once per visit at study center.
  Measures dynamic balance and fall risk by timing how long a person rises from a chair, walks 3 m, turns, returns and sits down.
6-Minute Walk Test (6MWT) | Baseline (t1), end of 3-week intervention (t3), and 3-week follow-up (t4) - performed once per visit at study center; distance in meters recorded.
  Assesses ambulatory endurance by recording the total distance walked (meters) in six minutes on a 12-m circuit.

CONTACTS AND LOCATIONS:
Locations (1):
- MEDIAN Rehab Center Wiesbaden Sonnenberg, Wiesbaden, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://saphenus-med.com/suralis/